CLINICAL TRIAL: NCT07099066
Title: Generation of Skin Fibroblast Banks, Urine-derived Cells and Biomarker Isolation From Patients With Amyotrophic Lateral Sclerosis (Als)
Brief Title: Generation of Cell Banks and Biomarker Isolation From Patients With Amyotrophic Lateral Sclerosis (ALS) (HCD-SLA)
Acronym: HCD-SLA
Status: Not yet recruiting | Type: Observational
Sponsor: Human Cell Design (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-A00776-43
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Cordocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALS patients
  Interventions: Other: sampling blood

INTERVENTIONS:
Other: sampling blood — 3 types of sampling : urine, skin and blood.

SUMMARY:
The aim of this research is to establish different cell banks from patients with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
The objective of this research is to:

* Create banks of skin fibroblasts from skin biopsy samples
* Create banks of urine-derived cells (UDCs) from urine samples
* Build a collection of blood samples to enable isolation of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years old;
* Subjects who have given their consent and signed an informed, free and express consent form;
* Subjects with diagnosed ALS;
* Subjects affiliated to or benefiting from a social security scheme.

Exclusion Criteria:

* Subjects with contraindications to the collection of biological samples (blood, skin, urine).
* Subjects undergoing treatment likely to affect hemostasis (anticoagulants, platelet anti-aggregants, etc.) in the month prior to inclusion and during the study;
* Subjects with hereditary or acquired haemostasis disorders;
* Subjects who have undergone physical treatment (radiotherapy, etc.) on the area to be biopsied in the last 6 months;
* Lidocaine-intolerant subjects;
* Subjects who have reached the age of majority and are subject to a protective measure or are unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS patients who are part of a cohort from the ALS Center of Toulouse University Hospital and are treated at that hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cell banking | 8 months
  Number of cell batches cryopreserved that meet predefined quality criteria (cell viability ≥ 80%, absence of mycoplasma). Data will be summarized as percentage of compliant batches over total batches produced.